CLINICAL TRIAL: NCT02752386
Title: Biofeedback Training to Control Pain Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Jamie Rhudy, Professor, University of Tulsa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TU1560
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biofeedback Training 1 (Experimental): Participants will receive brief training in relaxation and biofeedback to develop basic skills in relaxation/arousal reduction. Then they will receive instructions to relax and reduce arousal as they view graphical arousal feedback. Electric stimulations will be delivered throughout the biofeedback to provide pain relief when relaxation is achieved.
  Interventions: Behavioral: Biofeedback Training
- Biofeedback Training 2 (Active Comparator): Participants will receive brief training in relaxation and biofeedback to develop basic skills in relaxation/arousal reduction. Then they will receive instructions to relax and reduce arousal as they view graphical arousal feedback. Electric stimulations will be delivered throughout the biofeedback to provide a painful context in which to practice relaxing.
  Interventions: Behavioral: Biofeedback Training
- Biofeedback Training 3 (Active Comparator): Participants will receive brief training in relaxation and biofeedback to develop basic skills in relaxation/arousal reduction. Then they will receive instructions to relax and reduce arousal as they view graphical arousal feedback.
  Interventions: Behavioral: Biofeedback Training

INTERVENTIONS:
Behavioral: Biofeedback Training — Participants will received biofeedback training to reduce arousal and pain

SUMMARY:
The purpose of this study is to test whether a novel form of biofeedback training can help individuals regulate their pain more effectively.

DETAILED DESCRIPTION:
Relaxation is a low-cost treatment for managing pain with little or no side effects. The proposed study will use a novel biofeedback procedure to try to enhance the ability of relaxation to engage pain inhibition. Specifically, a biofeedback system will be used to provide training in conditioned pain regulation. The biofeedback system will monitor the trainee's level of sympathetic arousal and use it to control the intensity of painful stimulations delivered to the trainee during biofeedback. So when the trainee successfully relaxes (and reduced arousal), the intensity is lowered and produces pain relief. Efficacy of the training will be tested in a randomized controlled trial in which healthy, pain-free trainees are assigned to receive 3 training sessions or 3 sessions of a control procedure (2 other procedures will serve as controls; 3 groups total). The aim will be to assess whether the training results in inhibition of experimental pain and the nociceptive flexion reflex (NFR, a physiological marker of spinal pain signaling) to determine whether brain-to-spinal cord inhibitory circuits are engaged.

ELIGIBILITY:
Inclusion Criteria:

* healthy pain free individuals over the age of 18.

Exclusion Criteria:

* under 18 years of age (given the nature of the study)
* history of serious cardiovascular, neuroendocrine, or neurological disorders
* hypertension (due to a relationship between blood pressure and pain);5 4) history of chronic pain
* current opioid, antidepressant, or anxiolytic medication use
* psychosis or apparent cognitive impairment
* body mass index>35 (due to difficulty eliciting an NFR in persons with high adiposity)
* inability to understand and read English (questionnaires and consent form are in English)
* recent use of an over-the-counter pain medication (within the last 24 hours) or narcotic medication (within the last two weeks)
* history of panic attacks. No one will be excluded based on ethnic, racial, or gender characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in nociceptive flexion reflex threshold | Assessed at the beginning and end of each of the 3 biofeedback training days
  physiological marker of pain processing
Change in temporal summation of pain | Assessed at the beginning and end of each of the 3 biofeedback training days
  marker of pain facilitation (change in pain rating 0-100 that occurs in response to a mechanical stimulus series)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Rhudy, PhD, Principal Investigator — The University of Tulsa
Locations (1):
- University of Tulsa, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No